CLINICAL TRIAL: NCT06179355
Title: Comparison Between Manual Limbal Astigmatic Keratotomy and Femtosecond Laser-guided Limbal Astigmatic Keratotomy for Correction of Astigmatism More Than Three Diopters After Phacoemulsification
Brief Title: Limbal Astigmatic Keratotomy to Correct High Degrees of Astigmatism After Phacoemulsification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ashraf Rashwan, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1727367365
Record Dates: First submitted 2023-12-10; First posted 2023-12-21 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2023-10

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- manual Astigmatic Keratotomy (Experimental): manual limbal Astigmatic Keratotomy using a diamond knife group
  Interventions: Procedure: manual astigmatic keratotomy
- femtosecond laser Astigmatic Keratotomy (Experimental): Femtosecond laser-guided astigmatic keratotomy group
  Interventions: Procedure: femtosecond laser astigmatic keratotomy

INTERVENTIONS:
Procedure: manual astigmatic keratotomy — manual astigmatic keratotomy using a diamond knife
  Arms: manual Astigmatic Keratotomy
Procedure: femtosecond laser astigmatic keratotomy — astigmatic keratotomy using femtosecond lase
  Arms: femtosecond laser Astigmatic Keratotomy

SUMMARY:
Compare manually performed Astigmatic Keratotomy to femtosecond laser astigmatic keratotomy to manage corneal astigmatism more than three diopters after phacoemulsification.

DETAILED DESCRIPTION:
create circumferential corneal incisions, following the limbal curvature, at 1-1.5 mm anterior to the limbus, manually and by using femtosecond laser to correct corneal astigmatism more than three diopters after phacoemulsification.

ELIGIBILITY:
Inclusion Criteria:

* Possibility to have informed consent and attendance of all study visits.
* Patients who have undergone conventional phacoemulsification at least one month ago.
* Clear cornea.
* Astigmatism more than 0.5 diopters.

Exclusion Criteria:

* Corneal opacity.
* History of corneal surgery.
* Thin cornea.
* Astigmatism equal to or less than 0.5 diopters.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
astigmatism (Keratometric reading) | three month
  diopters of the astigmatism after the procedure measured by Pentacam

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Rashwan, MD, Principal Investigator — assiut univrsity
Locations (1):
- Faculty of Medicine, Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No